CLINICAL TRIAL: NCT03165435
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy of Subcutaneous Injections of the Active Targeted Immunotherapy CV-MG01 in Patients With Moderate to Severe Myasthenia Gravis.
Brief Title: A Study to Evaluate the Efficacy of CV-MG01 (Myasterix) in Myasthenia Gravis
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Not enough participating centres to complete recruitment in a timely manner.
Sponsor: CuraVac (Industry)
Collaborators: Aepodia (Industry); University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CV-0003; 2017-000323-27 (EudraCT Number)
Record Dates: First submitted 2017-05-17; First posted 2017-05-24 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Myasthenia Gravis, Generalized
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CV-MG01 (Experimental): The active targeted immunotherapy candidate, CV-MG01 comprises two short synthetic peptides separately conjugated to a carrier protein for the potential treatment of myasthenia gravis
  Interventions: Biological: CV-MG01
- Placebo (Placebo Comparator): Aluminium hydroxide adjuvant alone
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CV-MG01 — 3 consecutive subcutaneous injections of CV-MG01. The three injections are planned for each patient on Days 1, 29 (+/- 3 days) and 85 (+/- 7 days), respectively.
  Other Names: Myasterix
  Arms: CV-MG01
Biological: Placebo — 3 consecutive subcutaneous injections of placebo. The three injections are planned for each patient on Days 1, 29 (+/- 3 days) and 85 (+/- 7 days), respectively.
  Arms: Placebo

SUMMARY:
Study CV-0003 will be the second clinical trial administering CV-MG01 in humans. This will be a phase 2/3 proof-of-efficacy therapeutic confirmatory study following the proof-of-concept exploratory phase 1 study (CV-0002).

DETAILED DESCRIPTION:
The review of the clinical data accumulated so far in Study CV-0002 indicated that the safety and tolerability profile of CV-MG01 is considered very good, with positive immunogenicity results after the high dose regimen of CV-MG01. The preliminary results also show an indication of efficacy of CV-MG01, as based on the different scales and questionnaires results, all specific to MG disease. Therefore, it is proposed to investigate, in an appropriately designed, randomised, double-blind and powered study, the clinical efficacy of CV-MG01 in a larger cohort of MG patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Patient, with generalised myasthenia gravis (Grades 2, 3 and 4a) as per myasthenia gravis foundation of America (MGFA) classification system.
* Quantitative Myasthenia Gravis (QMG) score of 10 or greater at screening and baseline.
* Age of minimum 18, at the time of the consent form signature.
* Patient with documented positive antibodies to AChR in one of the available validated laboratory test.
* Patient may use corticosteroid treatment initiated for at least 3 months before screening, equivalent to a daily dose of 30mg prednisone as maximum, and stable (+/- 5mg change) at least 1 month before the screening and up to the first injection.
* Patient may use one or two immunosuppressive drugs (initiated for a least 6 months) with or without concomitant use of corticosteroid, providing that the dosage has been stable/unchanged for 3 months before the screening and up to the first injection.
* Venous access sufficient to allow blood sampling as per the protocol.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by the relevant Ethics Committee (EC) governing the site.

Exclusion Criteria:

* MG patients of Grade 5 based on myasthenia gravis foundation of America (MGFA) classification.
* Patients with history or presence of a primary or recurrent malignant disease including the presence or history of a thymoma.
* Thymectomy planned during Part A of the study period or performed within 1 year prior to the first dose of study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition not related to the treatment of MG, including human immunodeficiency virus (HIV) infection, or a family history of congenital or hereditary immunodeficiency.
* History or evidence of administration of immunoglobulins and/or any blood products within 3 months prior to the first dose of study drug, or a planned administration of immunoglobulins during the first 3 months of the study.
* History or evidence of rituximab treatment within 6 months prior to first dose of study.
* History or evidence of plasmapheresis within 3 months prior to the first dose of study, or a planned plasmapheresis during the first 3 months of the study.
* At high risk for aspiration.
* Pulmonary: forced vital capacity reduced to less than 70% of predicted capacity.
* History of severe allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History or evidence of Lambert-Eaton myasthenic syndrome, drug-induced myasthenia gravis, hereditary forms of myasthenic syndrome.
* History of relevant chronic degenerative, psychiatric, or neurological disorder other than MG.
* Severe hepatic, renal or cardiac insufficiency or uncontrolled hypertension
* Major congenital defects or serious chronic illness other than MG.
* Positive pregnancy test or desire to become pregnant during the study.
* Female patients of child-bearing potential that do not use a reliable and highly effective method of contraception (see Section 7.2 Contraception) at least one month before first injection, during the study and until the end of Part A.
* Any significant out-of-range Clinical Laboratory results considered as clinically significant and that prevent Subject's participation into the study according to Investigator's judgment.
* Previous completion or withdrawal from this study or study CV-0002.
* Sponsor employees or Investigator site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
* Any medical condition or concomitant medication that, in the opinion of the Investigator, might interfere with the subject's participation in the study, poses any added risk for the subject, or confounds the assessment of the subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy | 24 weeks
  To assess the efficacy of 3 subcutaneous injections of CV-MG01 compared to placebo, as measured by a decrease from baseline of the QMG total score at 24 weeks after the first injection (equivalent to 12 weeks after last injection).

SECONDARY OUTCOMES:
Safety (ohysical examens and laboratory tests) and local tolerance (FDA grading scale) | 24 weeks
  Evaluation of treatment emergent adverse events (TEAEs) including local injection site reactions (severity assessed with an overall grading scale following the FDA recommendation (FDA, CBER, September 2007)).
  General safety monitoring via physical examinations, vital signs (VS), ECG and standard laboratory tests (clinical chemistry, haematology and urinalysis).
Efficacy - Responder rate | 24 weeks
  Proportion of patients with improvement or worsening by ≥ 3 points in the QMG score at week 24 after the first injection in the active group compared to the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Mercelis, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital, Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Therapeutic Vaccines / Active Targeted Immunotherapies for Autoimmune Diseases — http://www.curavac.com